CLINICAL TRIAL: NCT03929757
Title: A Phase 2 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of a Heterologous 2-dose Vaccination Regimen Using Ad26.ZEBOV and MVA-BN®-Filo in Infants Aged 4-11 Months in Guinea and Sierra Leone
Brief Title: A Study of 2-dose Vaccination Regimen of Ad26.ZEBOV and MVA-BN-Filo in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Sierra Leone (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108617; VAC52150EBL2005 (Other: Janssen Vaccines & Prevention B.V.); 2021-001331-10 (EudraCT Number)
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — MenACWY

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Ad26.ZEBOV, MVA-BN-Filo (Experimental): Participants will be administered 0.5 mL of Ad26.ZEBOV vaccine (5*10^10 viral particles [vp]) on Day 1 by intramuscular (IM) injection followed by 0.5 mL of MVA-BN-Filo (1*10^8 infectious units [Inf U]) vaccine by IM injection on Day 57. Participants will also receive a dose of MenACWY at the 6-months post-dose-2 visit. Upon completion of the main study, participants in the extension phase who were originally randomized to the control arm will receive the same vaccine regimen as the participants in the Ad26.ZEBOV, MVA-BN-Filo arm of the main study.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: MenACWY
- Arm 2: MenACWY (Active Comparator): Participants will be administered 0.5 mL of MenACWY vaccine by IM injection on Day 1 and Day 57. Participants will also receive a dose of MenACWY at the 6-months post-dose-2 visit.
  Interventions: Biological: MenACWY

INTERVENTIONS:
Biological: Ad26.ZEBOV — Participants will receive 0.5 mL IM injection of Ad26.ZEBOV as first vaccination.
  Arms: Arm 1: Ad26.ZEBOV, MVA-BN-Filo
Biological: MVA-BN-Filo — Participants will receive 0.5 mL IM injection of MVA-BN-Filo as second vaccination.
  Arms: Arm 1: Ad26.ZEBOV, MVA-BN-Filo
Biological: MenACWY — Participants will receive 0.5 mL IM injection of MenACWY.

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of a heterologous 2-dose regimen utilizing Ad26.ZEBOV (first vaccination; Dose 1) and MVA-BN-Filo (second vaccination; Dose 2) administered intramuscularly (IM) on Days 1 and 57, respectively (Main Study) and also to provide the heterologous 2-dose vaccination regimen (Ad26.ZEBOV on Day 1 and MVABN-Filo on Day 57) to participants in the control arm of the main study (Extension Phase).

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) (preferably both if available or as per local requirements)/guardian must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for the study, and potential risks and benefits of the study, and are willing to allow their child to participate in the study
* Parent(s)/guardian are willing/able to ensure that their child adheres to the prohibitions and restrictions
* The parent(s)/guardian must be at or above the age of legal consent in the jurisdiction in which the study is taking place
* Infant must be healthy in the investigator's clinical judgment (and the parent(s)/guardian) on the basis of medical history, physical examination, vital signs and clinical laboratory tests performed at screening
* Infant has received all routine immunizations appropriate for his or her age at the time of enrollment as documented in the vaccination cards presented by the parent(s)/guardian. Participants are allowed to catch up on routine immunizations if needed (support for beneficial vaccines may be offered to participants)
* Extension Phase: Prior enrollment in the control arm of the main study and did not withdraw consent, and receipt of at least the first vaccination (Dose 1) in the main study

Exclusion Criteria:

* Having received any candidate or other Ebola vaccine
* History of Ebola virus disease (EVD), or prior exposure to Ebola virus, including travel to an area with a current Ebola outbreak less than 1 month prior to screening
* Having received any experimental candidate Ad26- or modified vaccinia ankara (MVA)-based vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines [for example, polysorbate 80, ethylenediaminetetraacetic acid (EDTA) or L-histidine for Ad26.ZEBOV vaccine; tris (hydroxymethyl)-amino methane (THAM) for MVA-BN-Filo vaccine and Neisseria meningitidis polysaccharide or tetanus toxoid for MenACWY]), including known allergy to chicken or egg proteins and aminoglycosides (gentamicin)
* Presence of acute illness (this does not include minor illnesses such as mild diarrhea or mild upper respiratory tract infection) or axillary temperature greater than or equal to (>=) 37.5 degree celsius on Day 1. Participants with such symptoms will be excluded from enrollment at that time but may be rescheduled for enrollment at a later date
* Extension Phase: Having received any candidate or other Ebola vaccine

Ages: 4 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (2):
- Centre National de Formation et de Recherche en Sante Rurale de Maferinyah, Conakry, Guinea
- College of Med and Allied Health Sciences, University of Sierra Leone, Freetown, Sierra Leone

REFERENCES:
- [Derived] Choi EM, Lacarra B, Afolabi MO, Ale BM, Baiden F, Betard C, Foster J, Hamze B, Schwimmer C, Manno D, D'Ortenzio E, Ishola D, Keita CM, Keshinro B, Njie Y, van Dijck W, Gaddah A, Anumendem D, Lowe B, Vatrinet R, Lawal BJ, Otieno GT, Samai M, Deen GF, Swaray IB, Kamara AB, Kamara MM, Diagne MA, Kowuor D, McLean C, Leigh B, Beavogui AH, Leyssen M, Luhn K, Robinson C, Douoguih M, Greenwood B, Thiebaut R, Watson-Jones D; EBOVAC-3/EBL2005 Study Team. Safety and immunogenicity of the two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen in infants: a phase 2, randomised, double-blind, active-controlled trial in Guinea and Sierra Leone. Lancet Glob Health. 2023 Nov;11(11):e1743-e1752. doi: 10.1016/S2214-109X(23)00410-2. PMID 37858585

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY: Healthy participants (infants) aged 4-11 months, were administered with 0.5 milliliter (mL) of adenovirus serotype 26 encoding the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) vaccine (5*10^10 viral particles [vp]) on Day 1 by intramuscular (IM) injection followed by 0.5 mL of Modified Vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo; 1*10^8 infectious units [Inf U]) vaccine by IM injection on Day 57. Participants also received a dose of World Health Organisation (WHO)-prequalified 0.5 mL of Meningococcal Group A, C, W135, and Y conjugate (MenACWY) vaccine by IM injection at the 6-months post-dose 2 visit, that is, Day 237.
- Main Study: MenACWY (Control Arm): Healthy participants were administered with 0.5 mL of MenACWY vaccine by IM injection on Day 1 and Day 57. Participants also received a dose of MenACWY vaccine by IM injection at the 6-months post-dose 2 visit, that is, Day 237.
- Extension Study: Ad26.ZEBOV + MVA-BN-Filo: Participants who were originally randomized to the control arm and who had not withdrawn during the main study entered the extension phase to receive 0.5 mL of Ad26.ZEBOV vaccine (5*10^10 vp) on Day 1 by IM injection followed by 0.5 mL of MVA-BN-Filo (1*10^8 Inf U) vaccine by IM injection on Day 57. Participants were also followed-up for safety until 28 days post-dose 2, that is, Day 85.
Period: Main Study: Up to Day 365
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm) | Extension Study: Ad26.ZEBOV + MVA-BN-Filo
Started | 75 | 33 | 0
Completed | 72 | 33 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by parent/guardian | 2 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Extension Study: Up to Extension Day 85
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm) | Extension Study: Ad26.ZEBOV + MVA-BN-Filo
Started | 0 | 0 | 26 (Only eligible participants entered extension study)
Completed | 0 | 0 | 25
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm) | Total
Number analyzed (Participants) | 75 | 33 | 108
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.7 (2.51) | 7.5 (2.66) | 7.6 (2.55)
Age, Customized [Count of Participants; unit: Participants]
  4 to <= 8 months | 43 | 19 | 62
  >8 to 11 months | 32 | 14 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 13 | 50
  Male | 38 | 20 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 19 | 55
  Unknown or Not Reported | 39 | 14 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 19 | 55
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 39 | 14 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  Guinea | 39 | 14 | 53
  Sierra Leone | 36 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants With Solicited Local and Systemic Adverse Events (AEs) up to 7 Days Post-dose 1
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site, were pre-defined local (at the injection site) AEs for which participant were specifically questioned and which were noted by participant in their diary for 7 days post vaccination. Solicited systemic events included fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills.
Time Frame: From dose 1 (Day 1) up to 7 days post-dose 1 (Day 8)
Population: The full analysis set included all participants with at least one study intervention administration documented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 75 | 33
Percentage of Participants
  Solicited Local AEs | 14.7 | 6.1
  Solicited Systemic AEs | 36.0 | 30.3

2. Primary Outcome: Main Study: Percentage of Participants With Solicited Local and Systemic AEs up to 7 Days Post-dose 2
Description: An AE is any untoward medical occurrence in a participants participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site, were pre-defined local (at the injection site) AEs for which participant were specifically questioned and which were noted by participant in their diary for 7 days post vaccination. Solicited systemic events included fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills.
Time Frame: From dose 2 (Day 57) up to 7 days post-dose 2 (Day 64)
Population: The full analysis set included all participants with at least one study intervention administration documented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 75 | 33
Percentage of Participants
  Solicited Local AEs | 9.3 | 9.1
  Solicited Systemic AEs | 29.3 | 33.3

3. Primary Outcome: Main Study: Percentage of Participants With Unsolicited AEs up to 28 Days Post-dose 1
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were events which were reported by the participant voluntarily or obtained by means of interviewing the participants in a nondirected manner.
Time Frame: From dose 1 (Day 1) up to 28 days post-dose 1 (Day 29)
Population: The full analysis set included all participants with at least one study intervention administration documented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 75 | 33
Percentage of Participants | 61.3 | 66.7

4. Primary Outcome: Main Study: Percentage of Participants With Unsolicited AEs up to 28 Days Post-dose 2
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were events which were reported by the participant voluntarily or obtained by means of interviewing the participant in a nondirected manner.
Time Frame: From dose 2 (Day 57) up to 28 days post-dose 2 (Day 85)
Population: The full analysis set included all participants with at least one study intervention administration documented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 75 | 33
Percentage of Participants | 57.3 | 72.7

5. Primary Outcome: Main Study: Percentage of Participants With Serious Adverse Events (SAEs) up to 6 Months Post Dose-2 on Day 57
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. A SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 6 months post dose-2 on Day 57 (Up to 8 months)
Population: The full analysis set included all participants with at least one study intervention administration documented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 75 | 33
Percentage of Participants | 13.3 | 12.1

6. Secondary Outcome: Main Study: Geometric Mean of Binding Antibody Levels Against the Ebola Virus Glycoprotein (EBOV GP)
Description: Geometric mean of binding antibody levels against the EBOV GP were reported.
Time Frame: 21 days post-dose 2 (Day 78)
Population: The per-protocol immunogenicity population included all randomized and vaccinated participants for whom immunogenicity data were available excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes (for example, missed Dose 2 vaccination, natural infections, etc.).
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/milliliter (EU/mL)
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 74 | 33
ELISA Units/milliliter (EU/mL) | 24309 [19695 to 30005] | NA [NA to NA] — Here, NA stands for data not available for geometric mean and confidence interval (CI) as the data was below lower limit of quantification (LLOQ) of 36.11 EU/mL.

7. Primary Outcome: Main Study: Percentage of Participants With SAEs Related to Study Intervention
Description: Percentage of participants with SAEs related to study intervention were reported. A SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Day 365
Population: The full analysis set included all participants with at least one study intervention administration documented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Ad26.ZEBOV + MVA-BN-Filo + MenACWY | Main Study: MenACWY (Control Arm)
Number analyzed (Participants) | 75 | 33
Percentage of Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Main study: Up to Day 365 ; Extension study: Up to extension Day 85
Description: The full analysis set included all participants with at least one study intervention administration documented.
Groups:
- Main Study: Ad26.ZEBOV+MVA-BN-Filo+MenACWY: Healthy participants (infants) aged 4-11 months, were administered with 0.5 milliliter (mL) of adenovirus serotype 26 encoding the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) vaccine (5*10^10 viral particles [vp]) on Day 1 by intramuscular (IM) injection followed by 0.5 mL of Modified Vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo; 1*10^8 infectious units [Inf U]) vaccine by IM injection on Day 57. Participants also received a dose of World Health Organisation (WHO)-prequalified 0.5 mL of Meningococcal Group A, C, W135, and Y conjugate (MenACWY) vaccine by IM injection at the 6-months post-dose 2 visit, that is, Day 237.
- Extension Study: Ad26.ZEBOV+MVA-BN-Filo: Participants who were originally randomized to the control arm and who had not withdrawn during the main study entered the extension phase to receive 0.5 mL of Ad26.ZEBOV vaccine (5*10^10 vp) on Day 1 by IM injection followed by 0.5 mL of MVA-BN-Filo (1*10^8 Inf U) vaccine by IM injection on Day 57. Participants were also followed-up for safety until 28 days post-dose 2, that is, Day 85.
Arm/Group | Main Study: Ad26.ZEBOV+MVA-BN-Filo+MenACWY | Main Study: MenACWY (Control Arm) | Extension Study: Ad26.ZEBOV+MVA-BN-Filo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/33 | 0/26
Serious Adverse Events (participants affected / at risk) | 10/75 | 4/33 | 0/26
Other Adverse Events (participants affected / at risk) | 58/75 | 26/33 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Ad26.ZEBOV+MVA-BN-Filo+MenACWY (N=75) | Main Study: MenACWY (Control Arm) (N=33) | Extension Study: Ad26.ZEBOV+MVA-BN-Filo (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Gastrointestinal Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Ad26.ZEBOV+MVA-BN-Filo+MenACWY (N=75) | Main Study: MenACWY (Control Arm) (N=33) | Extension Study: Ad26.ZEBOV+MVA-BN-Filo (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 6 (8) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 9 (10) | 7 (8) | 1 (1)
Conjunctivitis Bacterial (Infections and infestations) | 2 (3) | 2 (2) | 0 (0)
Furuncle (Infections and infestations) | 6 (6) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Gastrointestinal Candidiasis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Helminthic Infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Malaria (Infections and infestations) | 13 (15) | 9 (10) | 6 (9)
Nasopharyngitis (Infections and infestations) | 12 (13) | 6 (10) | 0 (0)
Oral Candidiasis (Infections and infestations) | 7 (7) | 3 (4) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 15 (19) | 9 (12) | 1 (2)
Rhinitis (Infections and infestations) | 10 (12) | 5 (5) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 8 (8) | 6 (9) | 3 (4)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03929757/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03929757/SAP_001.pdf